CLINICAL TRIAL: NCT04531865
Title: Efficacy and Safety of Mycophenolate Mofetil as Maintenance Therapy After Rituximab Treatment in Childhood-onset, Frequently-relapsing or Steroid-dependent Nephrotic Syndrome: a Multicenter Double-blind, Randomized, Placebo-controlled Trial
Brief Title: Randomized Trial Evaluating Mycophenolate Mofetil in Children With Nephrotic Syndrome After Rituximab Treatment
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: lack of funding
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Shanghai Children's Medical Center (Other); Shanghai Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FRSDRM
Record Dates: First submitted 2020-08-26; First posted 2020-08-31 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Frequently Relapsing Nephrotic Syndrome; Steroid-Dependent Nephrotic Syndrome
MeSH Terms: conditions — Nephrotic Syndrome | interventions — Rituximab; Mycophenolic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rituximab and Mycophenolate Mofetil (Experimental): First course Course Rituximab at Randomization. Addition of Maintenance Mycophenolate Mofetil from 4 Month onwards.
  Interventions: Drug: Rituximab; Drug: Mycophenolate Mofetil
- Rituximab Only (Placebo Comparator): First course Course Rituximab at Randomization. Addition of Maintenance Placebo tablets matching Mycophenolate mofetil from 4 Month onwards.
  Interventions: Drug: Rituximab; Drug: Placebo tablets matching Mycophenolate Mofetil

INTERVENTIONS:
Drug: Rituximab — Rituximab: 375 mg/m2 intravenously on day 0 and day 7
  Other Names: Rituximab Biosimilar HLX01
Drug: Mycophenolate Mofetil — Addition of Maintenance Mycophenolate Mofetil from 4 Month onwards. Dose: 20~30mg/kg/day，BID. Total duration : 8 months.
  Other Names: Mycophenolate Mofetil Dispersible tablets（CYCOPIN®）
  Arms: Rituximab and Mycophenolate Mofetil
Drug: Placebo tablets matching Mycophenolate Mofetil — Addition of Maintenance Placebo tablets matching Mycophenolate Mofetil from 4 Month onwards. Dose: 20~30mg/kg/day，BID. Total duration : 8 months.
  Arms: Rituximab Only

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of maintenance Mycophenolate Mofetil following single course of Rituximab in maintaining remission over 12 months among Children with frequently-relapsing or steroid-dependent nephrotic syndrome

DETAILED DESCRIPTION:
The results of multiple observational studies and randomized control trials have shown that Rituximab, a chimeric monoclonal antibody against the cluster of differentiation antigen 20 (CD20) antigen on B cells, is safe and effective for children with complicated steroid-dependent/ frequently-relapsing nephrotic syndrome (SDFRNS) without corticosteroid or immunosuppressive therapy. Single rituximab infusion has been shown to be efficacious for 6 to 12 months, the reported median relapse-free period was 9 months. Our previous study found that Mycophenolate mofetil can further improve the sustained remission time.

All patients will be treated with 2 doses of Rituximab 375 mg/m2 iv at time 0 and 7 days. Addition of Maintenance Mycophenolate Mofetil or placebo from 4 Month onwards. The expected duration of the follow-up is 12 months, consisting of 12 visits.

ELIGIBILITY:
Inclusion Criteria:

1. Children between 1 and 16 years with Frequently-relapsing or Steroid-dependent Nephrotic Syndrome
2. Estimated glomerular filtration rate (eGFR) ≥90 ml/min per 1.73 m2 at study entry.
3. Remission at study entry
4. Patients in whom ≥5 CD20-positive cells/μL are observed in the peripheral blood.
5. Parents willing to give informed written and audiovisual consent.

Exclusion Criteria:

1. Patients who have been diagnosed with nephritic- NS, such as immunoglobulin A(IgA) nephropathy, prior to assignment or in whom secondary NS is suspected.
2. Patients showing one of the following abnormal clinical laboratory values:

1) Leukocytes < 3000/μL. 2) Neutrophils < 1500/μL. 3) Platelets < 50,000/μL. 4) Alanine aminotransferase (ALT) > 2.5× upper limit of normal value. 5) Aspartate aminotransferase (AST) > 2.5× upper limit of normal value. 6) Positive for hepatitis B surface (HBs) antigen, HBs antibody, hepatitis B core (HBc) antibody, or hepatitis C virus (HCV) antibody. 7) Positive for HIV antibody.

3. Patients meeting one of the following infection criteria:

1) Presence or history of severe infections within 6 months prior to assignment.2) Presence or history of opportunistic infections within 6 months prior to assignment.3) Presence of active tuberculosis.4) Patients with a history of tuberculosis or in whom tuberculosis is suspected.5) Presence or history of active hepatitis B or hepatitis C or hepatitis B virus carrier.6) Presence of human immunodeficiency virus (HIV) infection.

4. Presence or history of angina pectoris, cardiac failure, myocardial infarction, or serious arrhythmia (findings observed under Grade 4 of the Common Terminology Criteria for Adverse Events (CTCAE)).

5. Presence or history of autoimmune diseases or vascular purpura.

6. Presence or history of malignant tumor.

7. History of organ transplantation.

8. History of drug allergies to methylprednisolone, acetaminophen, cetirizine, mycophenolate mofetil,rituximab, or any of the above drugs

9. Uncontrollable hypertension.

10. Having received a live vaccine within 4 weeks prior to enrollment.

11. Patients who do not agree with contraception during the study period.

12. Judged inappropriate for this study by the treating or study physicians.

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
1-year relapse-free survival rate | 1-year period after randomization
  The rate of no relapse within 1 year

SECONDARY OUTCOMES:
The concentration for MPA-area under curve(AUC) | At 48 weeks
  Blood concentrations of mycophenolic acid (MPA)
Proportion of patients with a relapse | 6 months period after randomization
  The proportion of patients with relapse
Time to relapse (days) | 1-year period after randomization
  Number of days from randomization to occurrence of first relapse
B-Cell Recovery Time | 1-year period after randomization
  Time to the first detection of CD19+ cells above 1% of total CD45+ lymphocytes after CD19+ cell depletion
Change in growth velocity | 1-year period after randomization
  The standard deviation scores (SDS) for height at 12th month minus that of randomization.
adverse events | 1-year period after randomization
  It is a binary variable (1/0). The varibale would be setted as "1" if any adverse events occours including early infusion termination, acute infusion reaction Infection, pulmonary fibrosis, encephalopathy, neutropenia. Adverse events graded according to Common Terminology Criteria For Adverse Events (NCI-CTCAE v4.03)

CONTACTS AND LOCATIONS:
Overall Officials: Xu Hong, PhD.MD., Principal Investigator — Children's Hospital of Fudan University
Locations (4):
- China (4):
  - Children's hospital of Fudan university, Shanghai, Shanghai Municipality
  - Shanghai Children's Hospital, Shanghai
  - Shanghai Children's Medical Center, Shanghai
  - Xinhua Hospital, Shanghai Jiaotong University School of Medicine, Shanghai